CLINICAL TRIAL: NCT04568447
Title: Pilot Study on the Effects of IMOOVE in Parkinson's Disease Patients
Acronym: IMOOVE-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 36/18
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; Imoove; Elispheric movement
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMOOVE (Experimental): Patients will undergo IMOOVE® treatment for 6 weeks, two times per week for a total of 12 treatments.
  Interventions: Device: IMOOVE

INTERVENTIONS:
Device: IMOOVE — Imoove® is a device dedicated to rehabilitation and fitness and has the capacity to increase muscle tenfold.

SUMMARY:
Parkinson's Disease (PD) is one of the most frequent causes of motor dysfunction in aging.

It is therefore important to use rehabilitative therapeutic approaches that may prevent the development of motor complications when possible.

Imoove® is a device dedicated to rehabilitation and fitness and has the capacity to increase muscle tenfold.

The project is focused on quantifying the efficacy of IMOOVE® as a treatment method for improving joint mobility, posture and autonomy in PD.

DETAILED DESCRIPTION:
The pathogenesis of PD-related postural abnormalities is probably multifactorial as well as widely indefinite, and this could compromise treatment choices and efficacy. In addition to dystonia and rigidity, proprioceptive and sensorimotor disintegration as well as peripheral degenerative processes (myopathy, skeletal and soft tissue changes) have been proposed as causative factors of abnormal trunk postures.

When the body is educated in the Elispheric® movement it relearns the original vertebral motion, and postural control necessary for any action by the body, the professional can then perform effective vertebral reeducation.

The Elispheric® movements are created by a motorised plate. This unique technology impulses the body through a centrifugal force in three planes. This force trains the body in its natural spirals.

The performance result is based on the fact that Imoove restores the all freedom of movement, strength, precision and it works on the basic skeletal posture.

It is an exploratory study, in order to verify if the project is adequate, to establish its feasibility and to obtain information that allows to determine the size of the sample of the definitive study, 30 consecutive PD outpatients will be recruited for the IMOOVE® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease (diagnosed according to UK Brain Bank Criteria);
* Age: 40-80
* Medical treatment for Parkinson's Disease must be stable for at least two weeks prior to inclusion, and during the study. During the study, the dosage of anti-parkinsonian drug treatment should not change, if it is not deemed necessary by the investigator.-

Exclusion Criteria:

* All the usual contraindications associated with physical medicine, rehabilitation and sport

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
MDS-UPDRS score | through study completion, an average of 1 year
  Change in the motor symptoms evaluated with the Movement Disorder Society Unified Parkinson's Disease Rating scale (MDS-UPDRS).
  Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum total UPDRS score is 199, indicating the worst possible disability from PD.

SECONDARY OUTCOMES:
EURO QOL-5D (EQ-5D) | through study completion, an average of 1 year
  Positive change in the quality of life score between 0-100 (from worst to better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: fabrizio stocchi, md phd, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Pisana, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
after the end of study
Supporting Information: Study Protocol, SAP
Time Frame: after the end of study
Access Criteria: request by email